CLINICAL TRIAL: NCT01172925
Title: Randomized Phase II Crossover Study of Tiotropium For Dyspnea in Advanced Non-Small Cell Lung Cancer
Brief Title: Study of a Tiotropium Inhaler For Shortness of Breath in Advanced Non-Small Cell Lung Cancer
Acronym: TIDAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, John Goffin, Associate Prof, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-TIDAL
Record Dates: First submitted 2010-07-22; First posted 2010-07-30 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: NSCLC; Dyspnea
Keywords: NSCLC; dyspnea; phase II; crossover; tiotropium
MeSH Terms: conditions — Dyspnea | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tiotropium (Experimental): Inhaler
  Interventions: Drug: Tiotropium
- Placebo (Placebo Comparator): Inhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium — Inhaler
  Arms: Tiotropium
Drug: Placebo — Inhaler
  Arms: Placebo

SUMMARY:
The feeling of shortness of breath is very common in lung cancer. It is uncomfortable for patients and upsetting for their family. Although drugs like morphine and oxygen can help some patients feel better, they don't help everybody, and they are not used in patients with early symptoms. More relief is needed for these patients. The investigators are studying a drug called tiotropium, which is used in emphysema. It is an inhaler that opens the airways to allow easier breathing. Every patient will get the drug but also a placebo, in a random (flip of a coin) order. They will get each for 2 weeks. The investigators will see if they feel better with the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven incurable stage IIIb or stage IV non-small cell lung cancer.
2. Dyspnea as defined by a score of 2 or higher on the 10-point Dyspnea Numeric Scale (Appendix 2).
3. New dyspnea or worsening dyspnea within the last 6 months per patient reporting.

Exclusion Criteria:

1. Age < 18.
2. An FEV1 / FVC ratio < 0.7 with an FEV1 of < 80% predicted post-bronchodilator.
3. Life expectancy < 3 months.
4. Significant worsening of dyspnea over the last week such that an acute cardiac or respiratory condition is considered likely (e.g. pneumonia, heart failure).
5. Myocardial infarction within the previous month.
6. Heart rate ≥ 120.
7. Active tuberculosis or tuberculosis receiving antibiotic therapy.
8. Current or previous use of ipratropium, tiotropium, or oxitropium (see Appendix 6).
9. Sensitivity to atropine.
10. Pre-existing diagnosis of asthma or moderate to severe Chronic Obstructive Pulmonary Disease
11. Use of beta-adrenergic bronchodilators more than once per week.
12. Use of experimental therapy with known cholinergic or adrenergic effects.
13. Uncontrolled glaucoma.
14. Urinary retention.
15. An active upper or lower respiratory infection or having taken antibiotics for any recent respiratory infection within 4 weeks.
16. Symptomatic pleural or pericardial effusion.
17. Evidence of reversible proximal endobronchial obstruction.
18. Oxygen saturation < 90%.
19. A hemoglobin of < 100 g/litre. Testing is to be within 4 weeks of randomization.
20. Calculated or urine creatinine clearance ≤ 50 mL/min (see Appendix 5 for calculation). Testing it to be within 4 weeks of randomization.
21. Weight loss > 10% of usual body weight within 6 months.
22. Known pregnancy or lactating.
23. Unable to independently fill out quality of life forms or give informed consent.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2010-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
12 question Cancer Dyspnea Scale | 6 weeks

SECONDARY OUTCOMES:
10 point Dyspnea numeric scale | 6 weeks
10 point Cough scale | 6 weeks
Forced Expiratory Volume 1 second (L/s) and Forced Vital Capacity (L) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Goffin, MD, Principal Investigator — Juravinski Cancer Centre and McMaster University
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada